CLINICAL TRIAL: NCT03606356
Title: Sustained onabotulinumtoxinA Therapeutic Benefits in Patients With Chronic Migraine Over 3 Years of Treatment. A
Brief Title: Sustained onabotulinumtoxinA Therapeutic Benefits in Patients With Chronic Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corfu Headache Clinic (Other)
Responsible Party: Principal Investigator, KONSTANTINOS SPINGOS, Konstantinos Spingos MD, Neurologist, Corfu Headache Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CorfuHC2
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — onabotulinum toxin A; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm, prospective multicentre, clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Onabotulinum toxin A — Cranial Subcutaneous Injections
  Other Names: Botox

SUMMARY:
To assess whether there is a sustained benefit and good safety with repeated onabotulinumtoxinA sessions in chronic migraine over more than three years of treatment.

We prospectively enrolled 65 chronic migraine patients, who were classified as responders after three sessions of onabotulinumtoxin A and were eligible to further continue treatment.

DETAILED DESCRIPTION:
Evidence on whether the therapeutic effect and good safety profile of onabotulinumtoxinA (Botox®) in chronic migraine (CM) patients is maintained over long term treatment is still limited. This study aims at assessing whether there is a sustained benefit and good safety with repeated onabotulinumtoxin A sessions in CM over more than three years of treatment.

This study prospectively enrolled 65 CM patients, who were classified as responders after three sessions of onabotulinumtoxinA and were eligible to further continue treatment. Data documenting longitudinal changes from the trimester after the third onabotulinumtoxinA administration (T1) to the trimester after completing two years of treatment (T2) and eventually to the trimester after completing three years of treatment (T3) in (i) mean number of monthly headache days (ii) migraine severity as expressed by the mean number of days with peak headache intensity of >4/10, and (iii) mean number of days with use of any acute headache medication, were prospectively collected from patients' headache diaries.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic migraine according to IHC-III with or without medication overuse.
* Responders defined as patients that after 3 sessions of treatment with onabutulinum toxin A, having experienced a ≥50% reduction in their average monthly migraine days

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Change in the mean number of monthly headaches | 3 years
  Change in the mean number of monthly headache days, from the third administration (months 10 to 12; T1) to the period after three years of treatment (months 37-39; T3)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vikelis M, Argyriou AA, Dermitzakis EV, Spingos KC, Mitsikostas DD. Onabotulinumtoxin-A treatment in Greek patients with chronic migraine. J Headache Pain. 2016 Dec;17(1):84. doi: 10.1186/s10194-016-0676-z. Epub 2016 Sep 17. PMID 27640152